CLINICAL TRIAL: NCT06436482
Title: Research of Endobronchial Optical Coherence Tomography in Pre-stage of Chronic Obstructive Pulmonary Disease
Brief Title: Research of Endobronchial Optical Coherence Tomography in Pre-COPD
Acronym: EBOCTIPCOPD
Status: Recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Guanghong Zhou, Attending physician, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPHGZ02
Record Dates: First submitted 2024-05-23; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Optical Coherence Tomography; Pulmonary Function
Keywords: Chronic Obstructive Pulmonary Disease; Optical Coherence Tomography; pre-stage
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: non-smoking with normal lung function, no other pulmonary diseases besides pulmonary nodule as indicated by chest computed tomography (CT).
  Interventions: Device: Optical Coherence Tomography
- Pre-stage of Chronic Obstructive Pulmonary Disease (Pre-COPD): Patients exhibit early pulmonary abnormalities, such as, CT scans show the presence of emphysema, bullae, and air trapping; pulmonary function manifested as preserved ratio impaired spirometry (PRISm). PRISm was defined as a normal ratio [the forced expiratory volume in one second (FEV1) / forced vital capacity (FVC) ≥ 0.7] after inhalation of a bronchodilator, but impaired ventilatory function [percentage of forced expiratory volume in the first second to the expected value (FEV1%) and/or percentage of FVC to the expected value (FVC%) < 80%], with concurrent structural changes in the lungs (such as emphysema) and/or physiological abnormalities (such as hyperinflation, decreased diffusion capacity, rapid decline in FEV1 )
  Interventions: Device: Optical Coherence Tomography
- Chronic Obstructive Pulmonary Disease (COPD): COPD was diagnosed based on GOLD guideline [1]; No acute exacerbations within 4 weeks; CT scans show no other pulmonary diseases besides COPD; pulmonary function test results were available from within the last 3 days. All COPD patients were treatment-naive except for those with at stage III-IV who received maintenance therapy
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — Placing the probe of OCT in RB10c through the working channel of bronchoscope for real time dynamic scanning and collecting OCT parameters from participants in different groups.

SUMMARY:
The pre-stage of Chronic Obstructive Pulmonary Disease (Pre-COPD) is challenging to diagnose. However, identifying Pre-COPD is a crucial step in the prevention and management of COPD. Endobronchial optical coherence tomography showed the value of diagnosis in Pre-COPD and COPD in previous researchs.

DETAILED DESCRIPTION:
We recruited COPD patients (stage I-II, n=15; stage III-IV, n= 15), Pre-COPD (n= 20) and healthy never-smokers (healthy human, n=21). Age,gender,BMI, smoking history, spirometry, chest computed tomography (CT), bronchoscopy and EB-OCT were performed. Inner luminal area (Ai) and airway wall area (Aw) of bronchi which inner perimeter was 10mm, 20mm and 30mm were measured using EB-OCT respectively. By analyzing and studying the above situation, we aim to discover the application value of OCT in Pre-COPD

ELIGIBILITY:
Inclusion Criteria:

* non-smoking with normal lung function, no other pulmonary diseases besides pulmonary nodule as indicated by chest computed tomography (CT).

Exclusion Criteria:

* (1) patients with contraindication of bronchoscopy, (2) patients who are participating in other clinical studies, (3) patients with poor compliance who are believed by the researchers to be unable to cooperate for the completion of the examination and follow-up, and (4) women who were pregnant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pre-COPD: Pre-COPD was diagnosed based on GOLD 2022; Patients exhibit early pulmonary abnormalities, such as, CT scans show the presence of emphysema, bullae, and air trapping; COPD: COPD was diagnosed based on GOLD guideline; No acute exacerbations within 4 weeks; CT scans show no other pulmonary diseases besides COPD; pulmonary function test results were available from within the last 3 days. All COPD patients were treatment-naive except for those with at stage III-IV who received maintenance therapy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Representative EB-OCT images of airway disorders | baseline
  Representative EB-OCT images(airway remodeling, mucosa thickening ) in CP，Pre-COPD and COPD
EB-OCT parameters in different stages of COPD | baseline
  Inner luminal area (Ai，mm) and airway wall area (Aw,mm2) of bronchi which inner perimeter was 10mm, 20mm and 30mm were measured using EB-OCT respectively.

SECONDARY OUTCOMES:
Baseline clinical characteristics | baseline
  Age（year）, gender(Male/female), smoking history(yes/no)
BMI（Kg/m2)） | baseline
pulmonary function test (FEV1 predicted %) | baseline
  Baseline clinical characteristics
FEV1/FVC ratio | baseline
MMEF 25/75 | baseline
  Baseline clinical characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Guanghong G Zhou, Master, Study Director — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided